CLINICAL TRIAL: NCT03391830
Title: Effects Of Combination Therapy Of Statin And Ascorbic Acid For Prevention Of Contrast-Induced Nephropathy. Randomised Controlled Study
Brief Title: Effects Of Combination Therapy Of Statin And Ascorbic Acid For Prevention Of Contrast-Induced Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Abdelwahab Hashem, Clinical Uro-oncology Fellow - Urology and Nephrology Center - Mansoura, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CN PREVENTION
Record Dates: First submitted 2017-12-30; First posted 2018-01-05 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2018-05

CONDITIONS: Contrast-induced Nephropathy; Statin; Ascorbic Acid; AKI

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atorvastatin-Ascorbic acid (Active Comparator): atorvastatin (80-mg loading dose given a mean 24 hours before procedure with another 40-mg dose approximately 2 hours before the procedure and for 3 days) plus ascorbic acid 500mg
  Interventions: Drug: Atorvastatin-Ascorbic acid
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin-Ascorbic acid — atorvastatin (80-mg loading dose given a mean 24 hours before procedure with another 40-mg dose approximately 2 hours before the procedure and for 3 days) plus ascorbic acid 500mg
  Arms: Atorvastatin-Ascorbic acid
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
To evaluate the benefit for statin use in prevention of of CI-AKI after computed tomography urogram (CTU).

ELIGIBILITY:
Inclusion Criteria:

* Planned computed tomography urogram (CTU)
* Statin naive, or not on statin treatment for at least 14 day

Exclusion Criteria:

* History of liver disease or elevated serum transaminases
* History of rhabdomyolysis or elevated creatinine kinase
* History of iodinated CM use within 14 days before randomization
* History of N-acetylcysteine, metformin or nonsteroidal anti-inflammatory drugs use within 48 hours of the procedure.
* History of hypersensitivity reaction to contrast media
* Pregnancy or lactation
* Acute renal failure
* End-stage renal disease requiring dialysis
* Cardiogenic shock or pulmonary edema
* Multiple myeloma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Contrast Induced-Acute Kidney Injury | 3 days
  Increase in serum creatinine ≥ 0.5 mg/dl or ≥ 25 % within 72 hours of contrast medium exposure.

SECONDARY OUTCOMES:
long-term Renal function by estimated GFR | 30 days
  measured in ml/min/1.73m2

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Othman, MD, Study Chair — Urology and nephrology center
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Aldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: No